CLINICAL TRIAL: NCT06712355
Title: A Phase III, Multisite, Double-blinded Randomized Trial of BNT327 in Combination With Chemotherapy (Etoposide/Carboplatin) Compared to Atezolizumab in Combination With Chemotherapy (Etoposide/Carboplatin) in Participants With First-line Extensive-stage Small-cell Lung Cancer
Brief Title: Safety and Efficacy of BNT327, an Investigational Therapy in Combination With Chemotherapy for Patients With Untreated Small-cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNT327-03; 2024-515765-34-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-11; First posted 2024-12-02 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Extensive-stage Small-cell Lung Cancer
Keywords: First-line ES-SCLC; SCLC; Immunotherapy in combination with chemotherapy; Untreated; Bispecific antibody; Programmed death-ligand 1 (PD-L1); Vascular endothelial growth factor (VEGF) A; Immunotherapy; Combination with other investigational agents; Pumitamig; BNT327; Check point inhibitor; Lung cancer; Etoposide; Carboplatin; Cisplatin
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — atezolizumab; Etoposide; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Stage 1 Control Arm - Atezolizumab + Etoposide + Carboplatin (Active Comparator)
  Interventions: Drug: Atezolizumab; Drug: Etoposide; Drug: Carboplatin (or cisplatin if carboplatin is not tolerated)
- Stage 1 Treatment Arm 1 - Pumitamig Dose 1 + Etoposide + Carboplatin (Experimental)
  Interventions: Drug: Pumitamig; Drug: Etoposide; Drug: Carboplatin (or cisplatin if carboplatin is not tolerated)
- Stage 1 Treatment Arm 2 - Pumitamig Dose 2 + Etoposide + Carboplatin (Experimental)
  Interventions: Drug: Pumitamig; Drug: Etoposide; Drug: Carboplatin (or cisplatin if carboplatin is not tolerated)
- Stage 2 Control Arm - Atezolizumab + Etoposide + Carboplatin (Active Comparator)
  Interventions: Drug: Atezolizumab; Drug: Etoposide; Drug: Carboplatin (or cisplatin if carboplatin is not tolerated)
- Stage 2 Treatment Arm - Pumitamig Dose 3 + Etoposide + Carboplatin (Experimental)
  Interventions: Drug: Pumitamig; Drug: Etoposide; Drug: Carboplatin (or cisplatin if carboplatin is not tolerated)

INTERVENTIONS:
Drug: Pumitamig — Intravenous infusion
  Other Names: BNT327; BMS-986545; PM8002
  Arms: Stage 1 Treatment Arm 1 - Pumitamig Dose 1 + Etoposide + Carboplatin; Stage 1 Treatment Arm 2 - Pumitamig Dose 2 + Etoposide + Carboplatin; Stage 2 Treatment Arm - Pumitamig Dose 3 + Etoposide + Carboplatin
Drug: Atezolizumab — Intravenous infusion
  Arms: Stage 1 Control Arm - Atezolizumab + Etoposide + Carboplatin; Stage 2 Control Arm - Atezolizumab + Etoposide + Carboplatin
Drug: Etoposide — Intravenous infusion and capsules
Drug: Carboplatin (or cisplatin if carboplatin is not tolerated) — Intravenous infusion

SUMMARY:
This is a Phase III, multisite, randomized, double-blinded study to investigate pumitamig (BNT327) combined with chemotherapy (etoposide/carboplatin) compared to atezolizumab combined with chemotherapy (etoposide/carboplatin) for the treatment of participants with previously untreated extensive-stage small-cell lung cancer (ES-SCLC).

DETAILED DESCRIPTION:
There are two stages in this study: Stage 1 will have two treatment arms and one control arm, and Stage 2 will have a treatment arm and a control arm. The control arms in Stages 1 and 2 are the same.

Each stage of the study consists of a screening period (up to 21 days), an induction period followed by a maintenance period (until confirmed disease progression, intolerable toxicity, participant withdrawal, study termination or up to 2 years [whichever occurs first]), and a follow-up (FU) period for all participants (2 safety FU visits and survival FU visits).

In Stage 1, eligible participants will be randomized (1:1:1) to the arms. In Stage 2, participants will then be randomized (1:1) to the arms. The randomization will be stratified based on the following factors:

1. Brain or liver metastases per investigator assessment (presence versus absence);
2. Smoking status (smoker versus never-smoker); and
3. Geography.

Participants will be allowed to switch to cisplatin if carboplatin is not tolerated at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed ES-SCLC (using the AJCC [American Joint Committee on Cancer] tumor node metastasis staging system combined with Veterans Administration Lung Study Group [VALG]'s two stage classification scheme). For AJCC tumor node metastasis staging system: AJCC 8th edition stage IV (T any, N any, M1a/b/c), or T3~4 for multiple lung nodules or tumor/nodule volume that cannot be encompassed in a tolerable radiotherapy plan.
* Have not had prior systemic therapy for ES-SCLC. However, participants with prior chemoradiotherapy for limited-stage-SCLC must have been treated with curative intent and had a treatment-free interval of at least 6 months after the last chemotherapy, radiotherapy, or chemoradiotherapy before diagnosis of ES-SCLC to be eligible.
* Have at least one measurable lesion as the targeted lesion based on RECIST v1.1. Lesions treated after prior local treatment (radiotherapy, ablation, interventional procedures, etc.) are generally not considered as target lesions. If the lesion with prior local treatment is the only targeted lesion, evidence-based radiology must be provided to demonstrate disease progression (the single bone metastasis or the single central nervous system metastasis should not be considered as a measurable lesion).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematologic and organ function as defined in the protocol.

Exclusion Criteria:

* Have histologically or cytologically confirmed SCLC with combined histologies.
* Have received any of the following therapies or drugs within the noted time intervals prior to study treatment:

  * Within 2 weeks: small molecule agents with half-life of <7 days; radiation outside the thoracic cavity including whole brain radiation. Of note, other local radiation for brain lesions (not whole brain) is allowed; local radiation for bone lesions is allowed. Palliative bone radiation or brain stereotactic radiosurgery would not require a washout period, but participants should recover from radiotherapy-related toxicity.
  * Within 4 weeks: radiation involving the thoracic cavity; small molecule targeted agents with half-life of ≥7 days; monoclonal antibodies, antibody-drug conjugates, radioimmunoconjugates, or T-cell or other cell-based therapies.
  * Have received prior treatment with anti-vascular endothelial growth factor (VEGF) monoclonal antibody, or programmed death (ligand)-1 (PD[L]-1)/VEGF bispecific antibody.
  * Have received systemic corticosteroids (at a dosage greater than 10 mg/day of prednisone or an equivalent dose of other corticosteroids) within 7 days prior to the initiation of study treatment. Note: local, intranasal, intraocular, intra-articular or inhaled corticosteroids, short-term use (≤7 days) of corticosteroids for prophylaxis (e.g., prevention of contrast agent allergy) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity reactions caused by exposure to allergens) are allowed.
* Have the following central nervous system metastases:

  * Participants with untreated brain metastases that are symptomatic or large (e.g., greater than 2 cm).
  * Participants with treated central nervous system (CNS) metastases who are not neurologically stable or on steroids (at a dosage greater than 10 mg/Day of prednisone or an equivalent dose of other corticosteroid) within 7 days before initiating study treatment of this study.
  * Participants with known leptomeningeal metastases.
* Have uncontrolled hypertension or poorly controlled diabetes prior to study treatment.
* Have a serious or non-healing wound, or (incompletely healed) bone fracture. This includes history of abdominal fistula, tracheoesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess for which an interval of 6 months must pass before study entry. In addition, the participant must have undergone correction (or spontaneous healing) of the perforation/fistula and/or the underlying process causing the fistula/perforation.
* Have a significant risk of hemorrhage (per investigator clinical judgment) as defined in the protocol.
* Have superior vena cava syndrome or symptoms of spinal cord compression that requires urgent medical intervention.

NOTE: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 46 months
  OS defined as the time from randomization to death from any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 46 months
  PFS defined as the time from randomization to first objective tumor progression (progressive disease per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1]), or death from any cause, whichever occurs first.
Objective response rate (ORR) | Up to approximately 46 months
  ORR defined as the proportion of participants in whom a complete response (CR) or partial response (PR) (based on investigator's assessment per RECIST v1.1) is observed as best overall response with confirmation.
Duration of response (DOR) | Up to approximately 46 months
  DOR defined as the time from onset of objective response (confirmed CR or PR based on investigator's assessment per RECIST v1.1) to first occurrence of objective tumor progression (progressive disease per RECIST v1.1) or death from any cause, whichever occurs first.
PFS rate based on investigator's assessment | At 6, 12, and 18 months
OS rate | At 6, 12, 18, and 24 months
Occurrence of treatment-emergent adverse events (TEAEs) including Grade ≥3, serious, and fatal TEAEs by relationship | From the first dose of study treatment to the 90-Day Follow-up Visit
  TEAEs graded according to (US) National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0
Occurrence of dose delay, infusion interruption and discontinuation of study treatment due to TEAEs (including related TEAEs) | From first to last dose of study treatment, i.e., up to 2 years
Change from baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality-of-Life Core 30 questionnaire (QLQ-C30) Global Health status/Quality-of-Life score (Items 29 and 30) | Up to approximately 46 months
  Global health status/QoL scale ranges in score from 0 to 100 with a high scale score representing a higher response level (e.g., high score for global health status/QoL is high QoL: high score for symptom scale/item is high symptomatology or problems).
Change from baseline in EORTC QLQ-C30 physical functioning | Up to approximately 46 months
  Physical functioning scale ranges in score from 0 to 100 with a high scale score representing a higher response level (e.g., high score for functional scale is high/healthy level of functioning).
Change from baseline in coughing scale of the EORTC Quality-of-Life-Lung cancer 29 questionnaire (QLQ-LC29) | Up to approximately 46 months
  Multi-item coughing scale ranges in score from 0 to 100 with a high score representing a high level of symptomatology or problems.
Change from baseline in shortness of breath scale of the EORTC QLQ-LC29 | Up to approximately 46 months
  Multi-item shortness of breath scale ranges in score from 0 to 100 with a high score representing a high level of symptomatology or problems.
Change from baseline in coughed up blood item of the EORTC QLQ-LC29 | Up to approximately 46 months
  Single item coughing up blood ranges in score from 0 to 100 with a high score representing a high level of symptomatology or problems.
Change from baseline in Functional Assessment of Cancer Therapy-General overall bother item (FACT-GP5). | Up to approximately 46 months
  The FACT-G - Item GP5 (Version 4) is a single-item summary measure of the overall impact of treatment toxicity, based upon its association with the number and degree of AEs in clinical studies, rated on a 5-point Likert scale ("not at all" to "very much") with a recall period of past 7 days. A high score represents high level of problems.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (107):
- United States (28):
  - Clermont Oncology Center, Clermont, Florida
  - Cancer Care Centers of Brevard, Inc, Palm Bay, Florida
  - Illinois Cancer Specialists, Niles, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc, Fort Wayne, Indiana
  - McFarland Clinic, Ames, Iowa
  - Helen G. Nassif Community Cancer Center, Cedar Rapids, Iowa
  - Baptist Health Hardin Cancer Center, Elizabethtown, Kentucky
  - Frederick Health Hospital- James M Stockman Cancer Institute, Frederick, Maryland
  - Beth Israel Lahey Health - Lahey Hospital & Medical Center (LHMC), Lahey Clinic Medical Center, Burlington, Massachusetts
  - Baptist Cancer Center, Southaven, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Hematology-Oncology (NHO), Lincoln, Nebraska
  - White Plains Hospital, White Plains, New York
  - Cleveland Clinic - Akron General Hematology & Oncology, Akron, Ohio
  - Cleveland Clinic Mercy Hospital Cancer Center, Canton, Ohio
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Cancer Center at Fairview Hospital, Moll Pavilion, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Cleveland Clinic - Hillcrest Hospital, Mayfield Heights, Ohio
  - St. Luke's Physician Group - St. Luke's Cancer Care Associates, Fountain Hill, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Millennium Research and Clinical Development, LLC, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Hematology Oncology Associates of Fredericksburg, Inc., Fredericksburg, Virginia
  - Shenandoah Oncology, Winchester, Virginia
- Australia (10):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Cancer Care Wollongong Pty Limited, Wollongong, New South Wales
  - Cairns Hospital, Cairns, Queensland
  - Icon Cancer Centre Kurralta Park, Kurralta Park, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Olivia Newton-John Cancer Wellness & Research centre, Heidelberg, Victoria
  - Western Health Sunshine Hospital, St Albans, Victoria
  - Cairns Hospital, Cairns
  - Royal North Shore Hospital, Saint Leonards
- China (16):
  - Jilin Cancer Hospital, Changchun, Jilin
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Chest Hospital,Capital Medical University, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Zhejiang Medical University, Zhejiang Cancer Hospital, Hangzhou
  - Jiamusi Cancer Hospital, Jiamusi
  - Shandong University - Jinan Central Hospital, Jinan
  - Shandong Cancer Hospital and Institute, Jinan
  - Linyi Cancer Hospital, Linyi
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Guangxi Tumour Hospital, Nanning
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Provincial Tumor Hospital (Shanxi Oncology Hospital), Taiyuan
  - The First Affiliated Hospital Of Wenzhou Medical University, Wenzhou
  - Xiangyang Central Hospital, Xiangyang
  - The First Affiliated Hospital of Henan Medical University, Xinxiang
- Japan (6):
  - Tokyo Metropolitan Komagome Hospital, Bunkyō City
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hospital Organization Himeji Medical Center, Himeji
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Sendai Kousei Hospital, Miyagi
  - Okayama University Hospital, Okayama
- South Korea (9):
  - Korea University Guro Hospital, Seoul, Guro-gu
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - The Catholic University Of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Gyeongsang National University Hospital (GNUH), Jinju, Gyeongsangnam-do
  - Gachon University Gil Medical Center, Incheon, Namdong-gu
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center (AMC), Seoul
  - Samsung Medical Center, Seoul
- Turkey (Türkiye) (21):
  - Acibadem Adana Hospital, Adana
  - Seyhan Medical Park Hospital, Adana
  - Baskent University Adana Turgut Noyan Application and Research Center, Adana
  - Ankara Etlik City Hospital, Ankara
  - Gulhane Training and Research Hospital, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara
  - Hacettepe University Medical Faculty Hospital, Ankara
  - Memorial Ankara Hospital, Ankara
  - Gazi University, Medical Faculty Hospital, Ankara
  - Liv Hospital Ankara, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Akdeniz University Hospital, Antalya
  - Trakya University Faculty of Medicine, Edirne
  - Koc Universitesi Hastanesi (Koc University Hospital), Istanbul
  - Medical Park Florya Hospital, Istanbul
  - Yeditepe University Kosuyolu Hospital, Istanbul
  - Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Medical Point Izmir Hospital, Izmir
  - Kocaeli University Medical Faculty Hospital, Kocaeli
  - Ankara University Medical Faculty Hospital, Mamak
  - Sakarya University Training and Research Hospital, Sakarya
- United Kingdom (17):
  - The Christie NHS Foundation Trust, Manchester, Lancashire
  - Royal Marsden Hospital (RMH) - Royal Marsden NHS Foundation Trust, Chelsea, London
  - Royal Marsden Hospital (Sutton) - Royal Marsden NHS Foundation Trust, Sutton, London
  - Huddersfield Royal Infirmary - Calderdale and Huddersfield NHS Foundation Trust, Huddersfield, North Yorkshire
  - Northern Centre for Cancer Care - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Northumberland
  - Nottingham University Hospitals NHS Trust - Nottingham City Hospital, Nottingham, Nottinghamshire
  - Churchill Hospital - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - Ninewells Hospital and Medical School - Tayside Health Board, Dundee, Scotland
  - Torbay and South Devon NHS Foundation Trust, Torquay, South Devon
  - Royal Stoke University Hospital - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire
  - Velindre NHS Trust, Velindre Cancer Centre, Cardiff, Wales
  - New Cross Hospital, Wolverhampton, West Midlands
  - Addenbrooke's Hospital - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Hull University Teaching Hospitals NHS Trust, Cottingham
  - Royal Devon and Exeter Hospital, Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - St James's University Hospital - Leeds Teaching Hospitals NHS Trust, Leeds
  - Royal Preston Hospital - Lancashire Teaching Hospitals NHS Foundation Trust, Preston

IPD SHARING:
Plan to Share IPD: No